CLINICAL TRIAL: NCT06771518
Title: Lung Microcytoma Extensive Disease: Prospective Study of Association of Thoraco-mediastinal Radiotherapy With Maintenance Immunotherapy Treatment With Atezolizumab
Brief Title: Association of Thoraco-mediastinal Radiotherapy With Maintenance Immunotherapy Treatment With Atezolizumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS1620/21
Record Dates: First submitted 2024-02-23; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: pharmacological interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thoracic radiotherapy-immunotherapy association in maintenance phase with atezolizumab (Experimental): Patients enrolled during the maintenance phase of chemoimmunotherapy treatment (standard of care) according to the IMPOWER 133 scheme which is divided as follows: 1) initial chemo-immunotherapy phase with IV treatment cycles with carboplatin AUC 5 day 1 and etoposide 100 mg/m2 days 1-3 q21 followed by a maintenance phase with immunotherapy (Atezolizumab day 1 1200 mg i.v. g1 of each cycle) until progression-toxicity.
  In association with immunotherapy, all patients will undergo treatment radiotherapy with 45 Gy in 15 fractions of 3 Gy administered 5 days a week on residual disease documented on CT-PET, dose 32.5Gy (2.16Gy for 15 fractions) on lymph node sites in response complete, equivalent to (EQD2 alpha beta 10) at 30 Gy in 3 fractions.
  Interventions: Radiation: Thoracic radiotherapy; Drug: Atezolizumab 1200 mg e.v. q21

INTERVENTIONS:
Radiation: Thoracic radiotherapy — Thoracic radiotherapy using 4D technique by irradiating the initial sites of disease (primary tumor and involved hilo-mediastinal lymph nodes). The treatments must be provided with the modulated intensity technique (IMRT or VMAT), treatments with conformal technique (3DCRT) are not permitted, where necessary, the Simultaneous Integrated Boost (SIB) technique can be used.
Drug: Atezolizumab 1200 mg e.v. q21 — Radiotherapy treatment associated with Atezolizumab 1200 mg i.v. q21 administered according to clinical practice

SUMMARY:
Investigate the role of consolidative radiotherapy treatment at the thoraco-mediastinal level in the patient suffering from lung microcytoma - extensive disease and treated with chemo-immunotherapy with atezolizumab, in association with maintenance therapy with atezolizumab.

DETAILED DESCRIPTION:
Prospective phase II study on patients affected by extensive-stage small cell lung cancer. The traditional treatment of lung microcytoma-extensive disease consists in platinum and etoposide-based chemotherapy. Radiotherapy of consolidation at the thoracic mediastinal level after chemotherapy may have an impact on survival and can be offered to patients in response to chemotherapy. Studies have recently shown that the addition of immunotherapy with atezolizumab to traditional chemotherapy improves survival compared to placebo. However, the use of consolidation radiotherapy was not permitted in the study thoracic level. Therefore the objective is to evaluate the efficacy and tolerance of the thoracic radiotherapy-immunotherapy association in the maintenance phase with atezolizumab of the treatment of lung microcytoma - extensive disease treated with chemo-immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of lung microcytoma;
* Age ≥18 years;
* Performance status according to ECOG 0-2;
* Extended disease at the time of first line oncological treatment;
* Initial staging and restaging after chemo-immunotherapy with CT, CT-PET FDG and brain MRI;
* In at least partial response (defined according to the Recist criteria [18]) after treatment chemoimmunotherapy according to the Impower 133 scheme;
* Haematological, respiratory toxicity ≤ G1, other toxicities ≤ G2 at the time of treatment radiotherapy;
* Pulmonary function tests at the time of radiotherapy treatment compatible with irradiation: FEV≥1.2 l or >40%, DLCO≥50%;
* Written informed consent.

Exclusion Criteria:

* Previous radiotherapy treatment at the thoraco-mediastinal level;
* In disease progression after chemo-immunotherapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of the association between radiotherapy and immunotherapy | 60 months
  The local recurrence rate of the disease at one year will be evaluated, with the aim of considering a % greater than 49.9% as unacceptable, assuming that with the experimental treatment object of this study a % of local recurrences of 30% can be achieved. We will therefore test the hypothesis of a local recurrence rate >50% vs the hypothesis of a local control <30%. Assuming a power of 80% and a one-sided significance level of 5%, it will be necessary to enroll 37 patients; if 13 or fewer local recurrences are observed, the study will be considered positive.

SECONDARY OUTCOMES:
Measuring the tolerability | 60 months
  The treatment will be considered feasible and non-toxic if severe toxicity values are found ≥ G3 similar or not higher than previous studies that used thoraco-mediastinal radiotherapy for consolidation after chemotherapy in the setting of small cell lung cancer - Extensive disease.
  In the present study, considering the use of modern radiotherapy techniques (IMRT or VMAT), the association of immunotherapy with thoracic radiotherapy in the maintenance phase will be considered feasible if an overall toxicity rate ≥ G3 < 20%, a respiratory toxicity grade ≥ G2 <10%, a respiratory toxicity grade ≥ G3 <5% is found. Toxicity will be evaluated according to the CTCAE V5.0 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy